CLINICAL TRIAL: NCT01792427
Title: Mortality in Non-cystic Fibrosis Bronchiectasis: a Long-term Cohort Analysis
Brief Title: Mortality in Non-cystic Fibrosis Bronchiectasis
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Dr. Lieven Dupont, prof. dr., Universitaire Ziekenhuizen KU Leuven
Other Study IDs: B51060; B32220084152 (Other: Belgium: Institutional Review Board)
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2013-02-20 (Estimated); Status verified 2013-02

CONDITIONS: Non-cystic Fibrosis Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
In this study we analyzed the overall survival for all newly diagnosed patients with non-cystic fibrosis bronchiectasis from June 2006 onwards. The investigators wanted to confirm the known risk factors such as age, gender, smoking history and Pseudomonas aeruginosa and evaluate the impact on survival of etiology, number of different bacteriological species in retrospective and prospective sputa, azithromycin use and presence/development of pulmonary hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically significant and radiologically proven bronchiectasis
* Chest CT scan confirming the presence of bronchiectatic lesions and had symptoms of chronic productive cough
* Bronchiectasis was deemed to be present if there was one or more of the following criteria: a bronchoarterial ratio greater than 1, lack of tapering of the bronchi and visualization of bronchi within 1 cm of costal or paravertebral pleura or abutting the mediastinal pleura

Exclusion Criteria:

* diagnosis of cystic fibrosis
* underlying tumoral problem causing the bronchiectatic lesions (postradiotherapy, secondary immunodeficiency due to chemotherapy or postinfectious due to tumoral obstruction)
* patients with asymptomatic traction bronchiectasis caused by interstitial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: non-cystic fibrosis bronchiectasis
Sampling Method: Non-Probability Sample
Enrollment: 253 (Actual)
Dates: Start 2006-06; Primary Completion 2012-10 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
overall survival | 6 years 4 months

SECONDARY OUTCOMES:
risk factor identification for NCFB | 6 years 4 months
  The investigators wanted to confirm the known risk factors such as age, gender, smoking history and Pseudomonas aeruginosa.

OTHER OUTCOMES:
Identify cause of death | 6 years 4 months
  If death occurred, the patient file was reassessed to identify cause of death.
risk factor identification for the survival of NCFB | 6 years 4 months
  The investigators will evaluate the impact of etiology, number of different bacteriological species in retrospective and prospective sputa, azithromycin use and presence/development of pulmonary hypertension on survival .

CONTACTS AND LOCATIONS:
Overall Officials: Pieter Goeminne, MD, Study Director — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium